CLINICAL TRIAL: NCT01197352
Title: Pilot Study of a Computer-driven Platform That Uses Text Messages to Collect Drinking Information and Deliver Personalized Motivational Messages to At-risk Young Adults
Brief Title: Pilot Study of a Text Message Platform to Reduce Risky Drinking in Young Adults
Acronym: PART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: PRO10040186
Record Dates: First submitted 2010-08-20; First posted 2010-09-09 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Alcohol Abuse; Alcohol Consumption; Drinking Behavior
Keywords: Alcohol; Abuse; Drinking; Behavior; Text; Computer
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Drinking Behavior; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Text message queries with feedback (Experimental): Weekly prompted queries about drinking behavior with personalized feedback.
  Interventions: Behavioral: Motivational and Normative Feedback
- Text message queries (Active Comparator): Weekly prompted queries about drinking behavior
  Interventions: Behavioral: Self-Awareness
- Control (No Intervention): Weekly text reminders to complete final (12 week) instruments

INTERVENTIONS:
Behavioral: Motivational and Normative Feedback — Weekly feedback based on their frequency and degree of at-risk drinking behavior using normative, educational and motivational feedback
  Arms: Text message queries with feedback
Behavioral: Self-Awareness — Weekly queries to raise awareness and allow self-reflection about drinking habits
  Arms: Text message queries

SUMMARY:
Young adults are in a critical period where they can be influenced to avoid a trajectory of high-risk drinking and harmful outcomes in the later adult years. The Emergency Department might offer a unique opportunity to reach young adults, if an easy to implement screening, brief intervention and referral to treatment was available. The investigators are investigating the feasibility and accuracy of ED-initiated and outpatient-continued assessment of drinking behavior in young adults using a computer-driven text messaging platform. Based on the subject's response to weekly assessments, the computer platform will send personalized motivational messages in real-time.

DETAILED DESCRIPTION:
Greater than 45% of young adults have heavy episodic drinking (HED; 5/4 drinks per occasion form men/women), resulting in significant health risks, including injury and death. Early identification and secondary prevention of HED using screening, brief interventions and referral to treatment (SBIRT) is advocated by the National Institute on Alcohol Abuse and Alcoholism (NIAAA) as a way to reduce injury and health consequences. Each day in the United States, there are over 2700 emergency department (ED) visits associated with alcohol, unfortunately, SBIRT is rarely performed in the ED due to time and training requirements. Our application seeks to solve this problem by integrating SBIRT into ED care through the use of ecological assessments with interventions. We will incorporate components of the NIAAA 2005 Clinicians Guide into automated weekly assessments (EA) and branching algorithms for personalized interventions (EA&I) delivered in real-time through mobile phone text messaging to young adults with a history of at-risk drinking behavior. We will assess the feasibility of EA&I to study young adults with a history of at-risk drinking and assess the variability in outcomes in patients undergoing EA&I, EA or standard care. We expect to find that this ED-initiated and outpatientcontinued platform will improve collection of drinking behavior, delivery of real-world motivational feedback and follow-up in young adults with at-risk drinking histories. We anticipate that short-term HED will be reduced in those subjects randomized to EA&I. We will use this information to support further studies with adequate power to show ED-initiated EA&I reduce long-term HED and its adverse consequences in young adults.

ELIGIBILITY:
Inclusion Criteria:

* 18-24 years
* English speaking
* Owns a personal phone with text messaging

Exclusion Criteria:

* Pregnant
* Prisoner
* Treated for alcohol dependence or abuse
* Treated for psychiatric disorder

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Ability of system to collect drinking information from young adults | 12 weeks
  We will report the proportion of weeks with completed drinking assessments in the EA and EA&I groups.

SECONDARY OUTCOMES:
Number of binge drinking episodes in subjects as a measure of safety and efficacy | 12 weeks
  We will compare the number of binge drinking episodes between subjects in the three groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center Emergency Department, Pittsburgh, Pennsylvania, United States